CLINICAL TRIAL: NCT02087462
Title: Electroacupuncture for Sciatica Due to Intervertebral Disc Displacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wu Xi, Principal Investigator, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011SZ0080
Record Dates: First submitted 2014-02-28; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Sciatica Due to Intervertebral Disc Disorder
Keywords: Sciatica; Electroacupuncture; Intervertebral disc displacement
MeSH Terms: conditions — Sciatica; Intervertebral Disc Displacement | interventions — Electroacupuncture; Traction; Diclofenac; Thiamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Electroacupuncture (EA) (Experimental): Use Electroacupuncture only
  Interventions: Other: Electroacupuncture (EA)
- EA + Traction (Other): Use electroacupuncture and traction together
  Interventions: Other: Electroacupuncture (EA); Other: Traction
- EA + Traction + Oral Medication (Other): Combine electroacupuncture, traction and oral medication (Voltaren and Vitamin B1) together for treatment
  Interventions: Other: Electroacupuncture (EA); Other: Traction; Drug: Voltaren; Drug: Vitamin B1

INTERVENTIONS:
Other: Electroacupuncture (EA) — Main acupoints: Da chang shu (BL25), Huan tiao (GB30), bilateral Jiaji point of attacked lumbar vertebra, Ashi points, modifying points according to different patterns.
  Electroacupuncture: choose the dilatational wave, frequency is 2Hz/100Hz, electric current ranges from 0.1mA to 1.0mA, 30 mins per time.
  Treatment frequency: 5 times per week in the first 2 weeks, 3 times per week in the 3rd and 4th week, 2 times per week in the 5th and 6th week.
  Duration: 6 weeks.
Other: Traction — An electric pelvis traction in supine position will be applied. The treatment frequency and duration are the same as EA.
  Arms: EA + Traction; EA + Traction + Oral Medication
Drug: Voltaren — Medication: 50 mg, twice per day
  Treatment frequency: In the first 2 weeks, take medicine for continuous 5 days with a 2-day interval each week; in the 3rd and 4th week, take medicine every 2 days, totally 3 times each week; in the 5th and 6th week, take medicine every 3 days, totally 2 times each week.
  Duration: 6 weeks.
  Other Names: Voltaren or Votalin.
  Arms: EA + Traction + Oral Medication
Drug: Vitamin B1 — Medication: 10mg, twice per day.
  Treatment frequency: In the first 2 weeks, take medicine for continuous 5 days with a 2-day interval each week; in the 3rd and 4th week, take medicine every 2 days, totally 3 times each week; in the 5th and 6th week, take medicine every 3 days, totally 2 times each week.
  Duration: 6 weeks.
  Other Names: Vitamin B1 or Thiamin or Thiamine or Aneurin
  Arms: EA + Traction + Oral Medication

SUMMARY:
This multicenter randomized controlled trial (RCT) will evaluate the therapeutic effectiveness and health-economics of electroacupuncture for sciatica due to intervertebral disc displacement in 3 compared groups: electroacupuncture, electroacupuncture plus traction, electroacupuncture plus traction and medication.

DETAILED DESCRIPTION:
This is a multicenter RCT with 3 groups to determine the effectiveness and health economic evaluation of the electroacupuncture for sciatica due to intervertebral disc displacement in a population of adults aged 18-65. 324 participants who meet the inclusion criteria will be randomly allocated into 3 different groups, namely electroacupuncture group, electroacupuncture & traction group, electroacupuncture & traction & oral medication group.

All participants will receive six-week treatment, the participants in electroacupuncture group will receive electroacupuncture only, electroacupuncture & traction group will receive both electroacupuncture and traction, and in electroacupuncture & traction & oral medication group all of the three therapies are adopted.

The statistical analysis will be conducted by a third party who is masked to the allocation of participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the clinical diagnosis of sciatica caused by intervertebral disc displacement;
* Male or female, aged 18-65;
* Have completed informed consent form.

Exclusion Criteria:

* Patients with sciatica caused by diseases such as piriformis syndrome, thickening of ligamentum flavus, acute lumbar strain, contusion, congenital spina bifid, lumbar and sacrum deformity, lumbar sacral vertebra joint disorder or proliferative osteoarthrosis;
* Patients with urinary and fecal incontinence caused by acute lumbar disc herniation, huge or central type lumbar disc herniation sufferer in need of surgery;
* Patients who fail to finish the basic treatment course, or have poor adherence;
* Patients having a poor state, particularly unconsciousness, psychopath, severe osteoporosis, concurrent infection or bleeding susceptibly, or accompany with primary diseases in cardiovascular, digestion or hemopoietic systems and viscera as kidney, liver;
* Pregnant or lactating women;
* Patients in other clinical research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) of Leg Pain | Change from baseline in VAS of Leg Pain at 6 weeks

SECONDARY OUTCOMES:
Visual Analog Scale(VAS) of Low Back Pain | Change from baseline in VAS of Low Back Pain at 6 weeks
Simplified McGill Pain Questionnaire (ST-MPQ) | Change from baseline in ST-MPQ at 6 weeks
Improved Roland Functional questionaire(RDQ) | Change from baseline in RDQ at 6 weeks
Likert Overall Recovery Self Rating Scale (7 points) | Change from baseline in Likert Overall Recovery Self Rating Scale at 6 weeks
The Medical Outcomes Study 36-Item Short -Form Health Survey Questionnaire (SF-36) | Change from baseline in SF-36 at 6 weeks
Sciatica Frequency and Bothersome Index (SFBI) | Change from baseline in SFBI at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xi Wu, A.P., Study Director — School of Acupunture& Tuina, Chengdu University of Traditional Chinese Medicine
Locations (1):
- Chengdu university of Traditonal Chinese Medcine, Chengdu, Sichuan, China